CLINICAL TRIAL: NCT03452761
Title: Effects of Exogenous Ketones in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Funding source: Pruvit Ventures, Inc (Unknown)
Responsible Party: Principal Investigator, Angelia Holland, Assistant Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 10414835
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Healthy Young Adults
Keywords: exogenous ketone salts; ketosis; safety; comprehensive metabolic panel; complete blood count; lipid panel; insulin
MeSH Terms: conditions — Ketosis; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, 2-groups (condition and placebo)
Who Masked: Participant, Investigator
Masking Description: Supplemental packets were not labeled except with the code A or B - placed by the supplement laboratory. PI notified of groups after completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Ketone Salts — Subjects will take 2 servings of ketone salts daily for 6 weeks
  Other Names: Exogenous Ketone Salts, Pruvit Keto OS

SUMMARY:
Exogenous ketone supplements in the form of beta-hydroxybutyrate can be utilized as an alternate energy source (in place of glucose) for all cells except red blood cells. Exogenous ketone administration has been shown to be beneficial in terms of reducing oxidative stress, improving neuronal energy supplies, and maintaining normal blood glucose levels. The purpose of this study is to determine the effects and safety of supplementing with exogenous ketones for 6-weeks in healthy college-aged males and females. The results of this proposed study will determine whether exogenous ketone supplementation can be useful in promoting better body composition, energy levels, and blood cholesterol, glucose, and insulin levels.

DETAILED DESCRIPTION:
A total of 22 subjects, male and female, were randomized to either a ketone salt group or a placebo group. Both the participants and investigators were blinded, as the supplements were coded by an external lab. Data was collected at baseline and again in 6-weeks. Participants consumed 2 servings of the assigned supplement daily for 6 weeks. Measures included body composition, blood pressure, questionnaires, blood work (comprehensive metabolic panel, complete blood count, and lipid panel), and a urinalysis. Also, blood ketone levels were assessed before and periodically after consuming the supplemental drink (30 and 60 minutes post drink). These measures were performed at both baseline and 6-weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no known conditions)

Exclusion Criteria:

* Chronic smoker Pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Blood health parameters | 6 weeks on the supplement
  Comprehensive Metabolic Panel
Blood health parameter | 6 weeks on the supplement
  Complete blood count
Blood health parameter | 6 weeks on the supplement
  Lipid Panel
Blood health parameter | 6 weeks on the supplement
  Insulin
Blood ketone levels | Baseline and 6 weeks after chronic consumption
  Blood ketones assessed 30- and 60 minutes after consuming the supplement
Cardiovascular | 6 weeks on the supplement
  Blood Pressure
Body Composition | 6 weeks on the supplement
  Skinfold measure
Body Composition | 6 weeks on the supplement
  Weight

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
All data will be deidentified